CLINICAL TRIAL: NCT04635670
Title: Effects of Probiotics and Fibers on Markers of Nephropathy, Inflammation and Endothelial Dysfunction in Persons With Type 1 Diabetes and Albuminuria
Brief Title: Effects of Probiotics and Fibers on Albuminuria in Persons With Type 1 Diabetes
Acronym: ProFOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H19070341
Record Dates: First submitted 2020-10-20; First posted 2020-11-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes; Nephropathy; Albuminuria; Diabetic Kidney Disease
Keywords: probiotics, dietary fibers
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Kidney Diseases; Albuminuria; Diabetic Nephropathies

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded, placebo controlled, crossover, single-centre study. A total of 46 participants will be randomly assigned into two groups of 23 to a sequence of treatment (active followed by placebo or vice versa). Allocation will be masked for both participants and investigators.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation will be masked for both participants and investigators. Only after completion of all study visits by all participants and after database lock the randomization code will be opened.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Soluble powder for oral use twice daily
  Interventions: Dietary Supplement: Placebo
- Active (Active Comparator): The investigational product is soluble powder for oral use of pre-/probiotic mix 3.0 g twice daily.
  Interventions: Dietary Supplement: Pro-/prebiotic Mix

INTERVENTIONS:
Dietary Supplement: Pro-/prebiotic Mix — Soluble powder for oral use of pre-/probiotic mix 3.0 g twice daily.
  Arms: Active
Dietary Supplement: Placebo — Soluble powder for oral use twice daily.
  Arms: Placebo

SUMMARY:
The primary objective is to assess the impact of three months' treatment with pre-/probiotic mix on markers of nephropathy and other comorbidity related to diabetes. A double blinded, randomized, placebo-controlled crossover, single-centre study including 46 patients with type 1 diabetes and albuminuria. The treatment period is 2 x 12 weeks with 6 weeks washout. The primary outcome is to evaluate the effect of pre-/probiotic mix on albuminuria.

DETAILED DESCRIPTION:
Recent data has pointed towards a link between gut microbiota and chronic kidney disease (CKD). It is hypothesized that defects in the intestinal barrier due to intestinal dysbiosis, a microbial imbalance in the intestines, allow bacterial toxins and other proinflammatory substances to pass and cause systemic inflammation that damages the endothelium. To reestablish the microbial symbiosis and thereby strengthening the gut barrier different treatments have been investigated. Fibers serve as substrate for the beneficial bacterial strains and probiotics are selected bacteria that exert a beneficial effect on the gut environment. It is hypothesized that a supplement of fructo-oligosaccharides and probiotics (Pre-/probiotic mix) will strengthen the gut barrier and thereby protect the endothelium and kidneys.

The aim of this study is to test whether af Pre-/probiotic mix, will have a beneficial impact on albuminuria in persons with type 1 diabetes and albuminuria.

46 patients with type 1 diabetes and albuminuria will be recruited from Steno Diabetes Center Copenhagen (SDCC) in accordance with the study in- and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Persons ≥ 18 years of age with a diagnosis of type 1 diabetes (age at onset <40 years; permanent insulin treatment initiated within 1 year of diagnosis)
2. Albuminuria: UACR > 30 mg/g (in ≥2 out 3 morning spot urine collections prior to randomization)
3. Participants must be on stable renin-angiotensin system blocking treatment 4 weeks before start of study drug and throughout study duration.
4. Able to understand the written participant information and give informed consent

Exclusion Criteria:

* 1. Non-diabetic kidney disease indicated by medical history and/or laboratory findings 2. Known inflammatory bowel disease (IBD) 3. IBD symptoms due to investigator's opinion 4. Known celiac disease 5. Existing ostomy, malabsorption, history of bowel resection or bariatric surgery.

  6. Heart valve replacement or history of endocarditis 7. Known rheumatic disorders treated with anti-inflammatory agents 8. Known hyperthyroidism or hypothyroidism 9. Active immunosuppressant therapy with systemic effect due to investigator's opinion 10. Current cancer treatment or within five years from baseline (except basal cell skin cancer or squamous cell skin cancer) 11. eGFR<15 ml/min/1.73m2, dialysis or kidney transplantation 12. Active antibiotic therapy until 30 days ahead of screening 13. Dietary supplements containing fibers (e.g. psyllium), probiotics or carotenoids until 30 days ahead of screening 14. The receipt of any investigational product 90 days prior to this trial 15. Unable to participate in study procedures 16. Any clinically significant disorder, except for conditions associated with type 1 diabetes, which in the Investigators opinion could interfere with the results of the trial 17. Pregnancy or lactation 18. Participation in another intervention study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Change in albuminuria based on urinary albumin-creatinine ratio (UACR) | 30 weeks. Samples will be collected before and after each og te two treatment periods.
  Three morning urine samples will be collected for assessment of UACR. The geometric mean of the 3 samples will be calculated.

SECONDARY OUTCOMES:
Change in kidney function (GFR as plasma clearance of 99mTc-DTPA) | 30 weeks. 99mTc-DTPA GFR will be performed after each of the two treatment periods.
  Renal function (GFR) and extracellular volume (ECV) will be assessed during 4 hours with the measurement plasma clearance of 99mTc-DTPA to provide accurate GFR measurement. A bolus of 0.5 mL Technetium-99m DTPA (approximately 10 MBq) is injected and blood samples are drawn at 0, 180, 200, 220 and 240 minutes after the injection. Urine is collected during the investigation. Plasma concentrations of 99mTc-DTPA at these time points are measured and used to calculate the plasma clearance of 99mTc-DTPA which approximates GFR.
Change in 24-hour blood pressure | 30 weeks. 24h BP will be performed after each of the two treatment periods.
  24-hours blood pressure will be measured using a standard cuff-based device (boso TM-2430 PC2) that measures the blood pressure every 15 minutes between 07 in the morning and 23 in the evening and every 30 minutes during the night.
Change in microcirculation evaluated by the GlycoCheck device | 30 weeks. GlycoCheck will be performed before and after each of the two treatment periods.
  GlycoCheck is a handheld video capillary microscope that measure glycocalyx thickness and sublingual capillary density under the tongue. The measurement will be performed by investigator and is a measure of the microcirculation damage. The distribution of the red blood cell column width at each capillary segment is used to calculate the perfused boundary region, which is the distance between the median and the outer edge of the red blood cell perfused lumen. The perfused boundary region reflects the thickness of the endothelial glycocalyx, based on the idea that loss of its integrity allows deeper penetration of the red blood cells into the gel-like layer covering the endothelial lining. Higher perfused boundary region, therefore, indicates thinner glycocalyx. The software also returns total and perfused capillary density in segments per millimeter square.
Change in endothelial dysfunction (von Willebrand factor, endothelin-1, ADMA, ICAM-1, VCAM-1 and E-selectin) | 30 weeks. Blood tests will be performed before and after each of the two treatment periods.
  Biomarkers drawn from blood will include markers of endothelial dysfunction (von Willebrand factor, endothelin-1, ADMA, ICAM-1, VCAM-1 and E-selectin),
Change in urinary markers of oxidative stress F2-isoprostanes and 8-oxodG | 30 weeks. Urine samples will be collected before and after each of the two treatment periods.
  Markers of oxidative stress (F2-isoprostanes and 8-oxodG) will be measured in urine by ELISA and multiplexing methods.
Change in intestinal inflammation measured by fecal calprotectin | 30 weeks. Fecal samples will be collected before and after each of the two treatment periods.
  Fecal samples will be collected for calprotectin analyses.
Change in biomarkers of intestinal permeability (LPS and zonulin) | 30 weeks. Blood tests will be performed before and after each of the two treatment periods.
  Biomarkers drawn from blood will include markers of intestinal permeability (LPS and zonulin)
Change in systemic inflammation (hs-TNT, TNF-alfa, IL6, IL8, IL1-beta, SAA, sICAM1, sICAM3 and suPAR) | 30 weeks. Blood tests will be performed before and after each of the two treatment periods.
  Biomarkers drawn from blood will include markers of inflammation (hs-TNT, TNF-alfa, IL6, IL8, IL1-beta, SAA, sICAM1, sICAM3, suPAR)
Change in tubular function (NGAL, KIM-1, Beta2microglobulin, hepatocellular growth factor and adiponectin) | 30 weeks. Urine samples will be collected before and after each of the two treatment periods.
  Markers of tubular kidney injury (NGAL, KIM-1, Beta2microglobulin, hepatocellular growth factor (HGF) and adiponectin) will be measured in urine by ELISA and multiplexing methods.
Change in autonomous neuropathy evaluated by VagusTM | 30 weeks. Vagus test will be performed before and after each of the two treatment periods.
  Autonomic nervous system function will be evaluated with the VagusTM device. The heart rate will be measured by 5-minute resting measures and in response to deep breathing, position change from lying to standing position and by exhaling through a mouthpiece against 40 mmHg of pressure (Valsalva maneuver).

OTHER OUTCOMES:
Change in concentration of microbial uremic toxins in the blood; hippuric acid, kynurenic acid, indoxyl sulfate and p-cresol sulfate | 30 weeks. Blood tests will be performed before and after each of the two treatment periods.
  Biomarkers will include markers of bacterial uremic toxins (hippuric acid, kynurenic acid, indoxyl sulfate and p-cresol sulfate).
Change in Gut microbiome characterization assessed by 16S RNA sequencing | 30 weeks. Fecal samples will be collected before and after each of the two treatment periods.
  Fecal samples will be collected at visit 2, 3, 4 and 5 for calprotectin and gut microbiome analyses. Feces is collected according to current standard operation procedures in order to characterize the gut microbiome. The fecal samples should be stored at -20 °C in the participants' freezer and be delivered to SDCC in the provided cooling bag no more than 48 hours after collection. At SDCC the samples will be stored at -80°C. The gut microbiome characterization is based on 16S rRNA gene sequencing. After standardized microbial DNA extraction, the microbial DNA will be subjected to sequencing, microbial gene analyses, taxonomy analyses including enterotypes known species and unknown meta-species and functional annotation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Proff, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No